CLINICAL TRIAL: NCT03054259
Title: A Feasibility Randomised Placebo-controlled Trial With Objective Outcome Measures to Evaluate the Efficacy of Biosimilar Rituximab in Musculoskeletal and Mucocutaneous Systemic Lupus Erythematosus
Brief Title: Rituximab Objective Outcome Measures Trial in SLE
Acronym: ROOTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RR15/197; 2015-002688-40 (EudraCT Number); 16/YH/0032 (Other: Research Ethics Committee Reference Number)
Record Dates: First submitted 2017-01-17; First posted 2017-02-15 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Systemic Lupus Erythematosus Arthritis
MeSH Terms: interventions — Rituximab; Methylprednisolone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 2 x 1000mg Rituximab and 100mg methylprednisolone
  Interventions: Drug: Rituximab; Drug: Methylprednisolone; Drug: Normal Saline
- Control (Placebo Comparator): 2 x 100mg methylprednisolone plus placebo
  Interventions: Drug: Methylprednisolone; Drug: Normal Saline

INTERVENTIONS:
Drug: Rituximab — 1000mg rituximab infusions on days 1 and 15 (monoclonal antibody)
  Arms: Intervention
Drug: Methylprednisolone — 100mg infusion on days 1 and 15
Drug: Normal Saline — 250ml infusion on days 1 and 15

SUMMARY:
This is a feasibility study to test a new trial design for an important drug in Systemic Lupus Erythematosus (SLE or "lupus").

SLE is an autoimmune disease. The immune system attacks the body's own tissues, any part of the body may be affected, but most commonly lupus causes a rash and arthritis, this affects patients' quality of life.

Lupus is usually treated with steroids or drugs that suppress the immune system. Although these help, many patients don't respond well enough and there is also concern for long term side effects. There is a new type of treatment called biologics. These target individual cells or molecules rather than the whole immune system and may be more effective with fewer side-effects. B cells are a part of the immune system that are known to play a role in lupus. There is already a biologic that removes these, called rituximab. In rheumatoid arthritis and vasculitis (similar to lupus), rituximab has been proven to be effective in clinical trials. However, in lupus clinical trials it did not seem to show any benefit. But many doctors and patients found that rituximab is effective, but the trials couldn't show this because of the way the drug's effects were measured. Therefore it is important that we test whether it truly is effective for lupus.

In this 6 month clinical study the investigators will look at lupus patients who have skin disease and arthritis as these are very common and randomise them to receive either rituximab or a placebo. Patients will have a careful clinical examination and undergo different methods to measure the effectiveness of the treatment. There are new versions to rituximab called "biosimilars". In this study biosimilar GP2013 will be used.

If this trial is successful a larger definitive study will be designed based on its results.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged at least 18 years old
* Active musculoskeletal SLE defined by inflammatory musculoskeletal pain with either clinical synovitis, ultrasound tenosynovitis or positive power Doppler in at least 1 joint
* No contraindication to the use of IV methylprednisolone, biosimilar rituximab, or any other required medications such as antipyretics and antihistamines
* Willing to use appropriate contraception if at risk of pregnancy
* Disease activity that is refractory to hydroxychoroquine, or patients unable to take hydroxychoroquine due to contra-indication or prior toxicity

Exclusion Criteria:

* • Severe "critical" SLE flare defined as: (i) BILAG 2004 A flare in CNS system; (ii) BILAG 2004 A flare in the renal system; or (iii) any other SLE manifestation requiring more immunosuppression than allowed within the protocol in the physician's opinion

  * Pregnancy
  * Breast Feeding
  * Receipt of daily oral glucocorticoids greater than 10mg prednisolone or equivalent at screening or within the previous 5 days, or change in glucocorticoid dose in the previous 5 days.
  * Receipt of intramuscular or intravenous glucocorticoids within the past 4 weeks
  * Receipt of intravenous immunoglobulin, plasma exchange or cyclophosphamide within the last 3 months
  * Rituximab within the past 18 months or other biologic therapies within the past 6 months
  * Active infections, including but not limited to the human immunodeficiency virus, hepatitis B (including prior infection as judged by positive Hepatitis B core antibody) or hepatitis C
  * Serum IgG below the lower limit of the local laboratory range
  * Receipt of a live attenuated vaccine within 3 months prior to study enrolment
  * History of cancer in the past 5 years except for squamous or basal cell carcinoma that has been completely excised or treated cervical carcinoma in situ
  * In female participants, known history of cervical dysplasia CIN Grade III cervical high-risk human papillomavirus or abnormal cervical cytology other than abnormal squamous cells of undetermined significance (ASCUS) within the past 3 years. The patient will be eligible after the condition has resolved (e.g., follow-up HPV test is negative or cervical abnormality has been effectively treated >1 year ago)
  * Planned surgery within the study period that is expected to require overnight hospital admission
  * Any other concomitant medical condition that, in the investigator's opinion, or after discussion with the CI, places the participant at risk by participating in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of trial considering adherence to protocol, completion of all assessments and visits | 26 weeks
  Overall feasibility of the trial will be judged based on the feasibility variables. It is acknowledged that this trial incorporates multiple inter-related aspects of design, with many possible modifications in trials derived from it. Hence these numbers will be used as a guide only and specific target values have not been defined.

SECONDARY OUTCOMES:
Proportion of patients achieving BILAG-based Composite Lupus Assessment (BICLA) | 16 weeks
  An assesment of clinical efficacy of treatment
Proportion of patients achieving SLEDAI responder Index (SRI) | 16 weeks
  An assesment of clinical efficacy of treatment
Number of serious adverse events | 26 weeks
  Safety assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Chapel Allerton Hospital- Leeds Institute for Rheumatic and Musculoskeletal Medicine, Leeds, West Yorkshire, United Kingdom